CLINICAL TRIAL: NCT06262230
Title: Feasibility and Effectiveness of Online Peer Companion Intervention on Children With Autism Spectrum Disorders
Brief Title: Feasibility and Effectiveness of OPCI on ASD Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University (Other)
Responsible Party: Principal Investigator, YinyinZang, Principal Investigator, Peking University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: OPCI on ASD Children
Record Dates: First submitted 2022-11-12; First posted 2024-02-15 (Actual); Last update posted 2024-02-15 (Actual); Status verified 2024-02

CONDITIONS: Autism Spectrum Disorder
Keywords: Autism Spectrum Disorder; Peer-Mediated Intervention
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Intervention Model Description: In this study, ordinary children will be paired with ASD children according to age, hobbies and other conditions
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- paired ASD and ordinary children (Experimental): In this prevent study, ordinary children will be paired with children with ASD based on ages, hobbies, and other aspects.
  Interventions: Behavioral: Online Inclusive Companionship Intervention

INTERVENTIONS:
Behavioral: Online Inclusive Companionship Intervention — After prior intervention, professionals will conduct a lecture for ordinary children, which includes basic knowledge of ASD and communication skills with ASD children. These ordinary children will be paired with ASD children then. The entire intervention including 12 sessions will last for 3 months. Researchers will prepare a series of themes that the ASD children could choose, and the ordinary children need to ask their paired ASD children what activities they want to choose before each session. Then, they will carry out this entertainment online together through Tencent WeMeet. A researcher will supervise online at the same time and record the communication through instant video. The Researcher will turn off the video and sound throughout the process and will not intervene in the conversation between the ASD children and ordinary children except for special circumstances.

SUMMARY:
The goal of this interventional study was to explore the feasibility and effectiveness of online peer companion intervention (OPCI) on the social abilities and mental health of ASD children. The main questions it aims to answer are:

1. What is the acceptability and adherence of OPCI;
2. Whether OPCI is effective on the social abilities and mental health of ASD children;
3. What impact does OPCI have on ordinary children and parents of both children?

DETAILED DESCRIPTION:
Autism Spectrum Disorder (ASD), as defined by the Diagnostic and Statistical Manual Fifth Edition of the American Psychiatric Association (DSM 5), is a neurodevelopmental disorder associated with symptoms that include "persistent deficits in social communication and social interaction across multiple contexts" and "restricted, repetitive patterns of behavior, interests, or activities." The education of children with ASD is a critical topic that has attracted widespread attention around the world. The mainstream education model has gradually shifted from the traditional education that separates special groups from the general population to a new model named inclusive education. Inclusive education was formally proposed in the Salamanca Declaration promulgated by the World Conference on Education for All in 1994, which was organized by the United Nations Educational, Scientific and Cultural Organization. The so-called inclusive education is an educational concept of special education, which means that children with disabilities could enter common classes for non-differentiated learning through different levels of educational design and adjustment. However, due to problems such as teachers' competence and public awareness, it is difficult to popularize and popularize inclusive education in schools in China. According to the data of the "White Paper on the Investigation of Family Situation of Autism in China", although over 70% of the people said they were not afraid of contacting autistic patients, over 80% of the people said they would accept and help autistic patients. As a result of the insufficient understanding of autism, only about 10% of children with ASD could enter ordinary schools. Based on this actual condition, the inclusive education of ASD children in China is mainly led by social organizations and guides ordinary children and ASD children to carry out activities together by stimulating ordinary children's curiosity and sympathy for the population of ASD children.

The effectiveness of the inclusive education model through peer-to-peer entertainment has also received preliminary empirical support. A study by Zercher et al. (2001) showed that, after training, typically developing groups of children aged 5, 9, and 11 were able to effectively promote activities in comprehensive playgroups involving children with ASD, whereas During this process, the characteristics of children with ASD, such as attention and verbal expression, were significantly improved. The results also showed that such increases were maintained in the unassisted group. Some studies have also shown that this form of inclusive education not only has a significant effect on the improvement of symptoms of ASD children, but also has a positive impact on the mental health of ordinary children, and can improve their self-efficacy and life satisfaction.

In recent years, the COVID-19 epidemic has had a huge impact on the world. To ensure the safety and health of children, inclusive education cannot be carried out offline. Fortunately, online inclusive education has achieved initial development. Furthermore, the development of online inclusive education could balance the differences in mental health resources between different regions. However, the feasibility and effectiveness of online inclusive education have yet to be clarified. Based on this background, this study will take ASD children and ordinary children of the same age population as participants. this present study aims to preliminarily clarify the feasibility and effectiveness of one-to-one online communication and peer-to-peer entertainment.

This present study will explore the feasibility and effectiveness of online peer companion intervention (OPCI) for children with ASD. Compared to traditional offline education and interventions for ASD children, this online intervention has higher convenience and lower cost advantages. At the same time, OPCI is also conducive to balancing the differences in mental health resources, so that more children with ASD from underdeveloped regions could have better interventions. Furthermore, in addition to improving social skills and mental health, peer participation in OPCI has the potential to promote the development of the social networks of children with ASD.

ELIGIBILITY:
Inclusion Criteria of ASD Children:

* 7-15 years old and diagnosed as mild ASD;
* Basic ability to speak independently and fluently communicate with peers;
* Could use mobile phones, tablets, computers, or other electronic devices for this online intervention.

Exclusion Criteria of ASD Children:

* Diagnosed as moderate or severe ASD;
* Unable or unwilling to communicate with peers independently
* No phones or other alternative electronic devices for the intervention

Inclusion Criteria of Ordinary Children:

* 9-18 years old with normal development, no diagnosis of ASD, learning disabilities, ADHD, and other mental disorders;
* Lively and outgoing, able to assume the role of topic organizer in communication with peers;
* Could use mobile phones, tablets, computers, or other electronic devices for this online intervention.

Exclusion Criteria of Ordinary Children

* Diagnosis of ASD or other neurodevelopmental and mental disorders;
* Introverted or unwilling to play with peer ASD children
* No phones or other alternative electronic devices for the intervention

Ages: 7 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2022-11-20 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2023-10-31 (Actual)

PRIMARY OUTCOMES:
Social Behavior of ASD Children | Pre-test, two process measurements (after 6th and 9th session, respectively), post-test, and follow-up (1, 2, 3 and 6 months after the intervention)
  We explored the effectiveness of OPCI on the social behavior of ASD participants through some parent-report scales, including the Social Responsiveness Scale (SRS) and the Strengths and Difficulties Questionnaire (SDQ).
Mental Health of ASD Children | Pre-test, two process measurements (after 6th and 9th session, respectively), post-test, and follow-up (1, 2, 3 and 6 months after the intervention)
  We explored the effectiveness of OPCI on the mental health of ASD participants through the parent-report 25-item Revised Child Anxiety and Depression Scale (RCADS).
Intervention Process Screen Recording Coding | each session
  We coded the screen recording of interventions to explore the effectiveness and influencing factors of OPCI. Videos for each dyad will be conducted by a trained undergraduate student. This work will be carried out under the guidance and supervision of a professional clinical psychologist.
Symptom Severity | Pre-test, two process measurements (after 6th and 9th session, respectively), post-test, and follow-up (1, 2, 3 and 6 months after the intervention)
  We explored the effectiveness of OPCI on the ASD symptoms through the Autism Behavior Checklist (ABC), which is a parent-report scale

SECONDARY OUTCOMES:
Mental Health of Ordinary Children | Pre-test, two process measurements (after 6th and 9th session, respectively), post-test, and follow-up (1, 2, 3 and 6 months after the intervention) or only measure at pre-test, post-test and follow-up.
  We explored the effectiveness of OPCI on the mental health of ordinary children participants through some self-report and parent-report scales, including the 25-item Revised Child Anxiety and Depression Scale (RCADS), Perceived Stress Scale (PSS), Self Acceptance Questionnaire (SAQ), Connor-Davidson resilience scale (CD-RISC), and so on.
Social Ability of Ordinary Children | Pre-test, two process measurements (after 6th and 9th session, respectively), post-test, and follow-up (1, 2, 3 and 6 months after the intervention)
  We explored the effectiveness of OPCI on the social ability of ordinary children participants through self-report and parent-report Social Skills Rating Systems (SSRS)
Mental Health of Parents | Pre-test, two process measurements (after 6th and 9th session, respectively), post-test, and follow-up (1, 2, 3 and 6 months after the intervention) or only measure at pre-test, post-test and follow-up.
  We explored the effectiveness of OPCI on the mental health of both children's parents through some self-report scales, including the General Anxiety Disorder Scale-7 (GAD-7), Patient Health Questionnaire-9 (PHQ-9), Perceived Stress Scale-4 (PSS-4), Self Acceptance Questionnaire (SAQ), Connor-Davidson resilience scale (CD-RISC), and so on.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No
Since this study would include ASD children, we didn't plan to share IPD to protect the participants in this study

REFERENCES:
- [Background] Chen YL, Schneider M, Patten K. Exploring interpersonal and environmental factors of autistic adolescents' peer engagement in integrated education. Autism. 2022 Jul;26(5):1255-1266. doi: 10.1177/13623613211046158. Epub 2021 Sep 18. PMID 34541934
- [Result] Zercher C, Hunt P, Schuler A, Webster J. Increasing joint attention, play and language through peer supported play. Autism. 2001 Dec;5(4):374-98. doi: 10.1177/1362361301005004004. PMID 11777255
- [Result] Jones, V. (2007). 'I felt like I did something good'-The impact on mainstream pupils of a peer tutoring programme for children with autism. British Journal of Special Education, 34(1), 3-9. https://doi.org/10.1111/j.1467-8578.2007.00447.x